CLINICAL TRIAL: NCT05669534
Title: Optimizing Evidence-based HIV Prevention Targeting People Who Inject Drugs on PrEP
Acronym: MOST
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Michael Copenhaver, Professor, University of Connecticut
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: H22-0121
Record Dates: First submitted 2022-12-05; First posted 2023-01-03 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Hiv; Opioid Use Disorder
Keywords: people who inject drugs; HIV; cognitive dysfunction; pre-exposure prophylaxis; multiphase optimization strategy; medication for opioid use disorder; opioid use disorder
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Opioid-Related Disorders; Cognitive Dysfunction | interventions — Pre-Exposure Prophylaxis; Post-Exposure Prophylaxis

STUDY DESIGN:
Intervention Model Description: Multiphase Optimization Strategy
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (16):
- Condition 1 (Active Comparator): Standard CHRP Intervention Components
  Interventions: Behavioral: community-friendly health recovery program; Drug: Pre-Exposure Prophylaxis and Post-Exposure Prophylaxis
- Condition 2 (Experimental): Standard CHRP Intervention Components and Information Processing Components
  Interventions: Behavioral: community-friendly health recovery program; Drug: Pre-Exposure Prophylaxis and Post-Exposure Prophylaxis
- Condition 3 (Experimental): Standard CHRP Intervention Components and Memory Components
  Interventions: Behavioral: community-friendly health recovery program; Drug: Pre-Exposure Prophylaxis and Post-Exposure Prophylaxis
- Condition 4 (Experimental): Standard CHRP Intervention Components, Information Processing Components, and Memory Components
  Interventions: Behavioral: community-friendly health recovery program; Drug: Pre-Exposure Prophylaxis and Post-Exposure Prophylaxis
- Condition 5 (Experimental): Standard CHRP Intervention Components, Executive Functioning Components
  Interventions: Behavioral: community-friendly health recovery program; Drug: Pre-Exposure Prophylaxis and Post-Exposure Prophylaxis
- Condition 6 (Experimental): Standard CHRP Intervention Components, Information Processing Components, and Executive Functioning Components
  Interventions: Behavioral: community-friendly health recovery program; Drug: Pre-Exposure Prophylaxis and Post-Exposure Prophylaxis
- Condition 7 (Experimental): Standard CHRP Intervention Components, Memory Components, and Executive Functioning Components
  Interventions: Behavioral: community-friendly health recovery program; Drug: Pre-Exposure Prophylaxis and Post-Exposure Prophylaxis
- Condition 8 (Experimental): Standard CHRP Intervention Components, Information Processing Components, Memory Components, and Executive Functioning Components
  Interventions: Behavioral: community-friendly health recovery program; Drug: Pre-Exposure Prophylaxis and Post-Exposure Prophylaxis
- Condition 9 (Experimental): Standard CHRP Intervention Components and Attention Components
  Interventions: Behavioral: community-friendly health recovery program; Drug: Pre-Exposure Prophylaxis and Post-Exposure Prophylaxis
- Condition 10 (Experimental): Standard CHRP Intervention Components, Information Processing Components, and Attention Components
  Interventions: Behavioral: community-friendly health recovery program; Drug: Pre-Exposure Prophylaxis and Post-Exposure Prophylaxis
- Condition 11 (Experimental): Standard CHRP Intervention Components, Memory Components, and Attention Components
  Interventions: Behavioral: community-friendly health recovery program; Drug: Pre-Exposure Prophylaxis and Post-Exposure Prophylaxis
- Condition 12 (Experimental): Standard CHRP Intervention Components, Information Processing Components, Memory Components, and Attention Components
  Interventions: Behavioral: community-friendly health recovery program; Drug: Pre-Exposure Prophylaxis and Post-Exposure Prophylaxis
- Condition 13 (Experimental): Standard CHRP Intervention Components, Executive Functioning Components, and Attention Components
  Interventions: Behavioral: community-friendly health recovery program; Drug: Pre-Exposure Prophylaxis and Post-Exposure Prophylaxis
- Condition 14 (Experimental): Standard CHRP Intervention Components, Executive Functioning Components, Attention Components, and Information Processing Components
  Interventions: Behavioral: community-friendly health recovery program; Drug: Pre-Exposure Prophylaxis and Post-Exposure Prophylaxis
- Condition 15 (Experimental): Standard CHRP Intervention Components, Executive Functioning Components, Attention Components, and Information Processing Components
  Interventions: Behavioral: community-friendly health recovery program; Drug: Pre-Exposure Prophylaxis and Post-Exposure Prophylaxis
- Condition 16 (Experimental): Standard CHRP Intervention Components, Executive Functioning Components, Attention Components, Information Processing Components, and Memory Components
  Interventions: Behavioral: community-friendly health recovery program; Drug: Pre-Exposure Prophylaxis and Post-Exposure Prophylaxis

INTERVENTIONS:
Behavioral: community-friendly health recovery program — Participants will receive 4 weekly 45 minute sessions HIV prevention sessions.
  Other Names: CHRP
Drug: Pre-Exposure Prophylaxis and Post-Exposure Prophylaxis — Participants will be prescribed Pre-exposure prophylaxis (PrEP) is a biomedical intervention.
  Other Names: PrEP

SUMMARY:
The investigators will conduct an optimization trial among N=256 PWID newly started on medication for opioid use disorder and Pre-Exposure Prophylaxis (PrEP) to assess the performance of four intervention components (Attention, Executive Functioning, Memory, and Information Processing) aimed at enhancing the ability of PWID on MOUD to process and utilize HIV prevention content, leading to improvements in HIV prevention information, motivation, behavioral skills, and behaviors (IMB).

DETAILED DESCRIPTION:
Participants will be randomized to one of 16 conditions. In addition to receiving the Core Components of the CHRP behavioral intervention, participants will receive one of the sixteen combinations of four compensatory components that show promise in terms of enhancing the ability to process and utilize HIV prevention content (see conceptual figure above), and that are not currently part of CHRP. The Attention Component includes: (a) Increasing frequency of sessions (more than once per week); (b) Distributed practice (spreading out information across sessions); (c) More structured sessions (well-organized objectives shared with patients); (d) Introducing new information during closure (foreshadow content of next session). The Executive Function Component includes the following strategies: (a) Associating behavior with situational cues (anticipate risky situations); (b) Linking actions to a triggering cue (storytelling techniques using imagery); (c) Planning (identify and organize steps required to meet goal) and (d) Valuing future events (recognize the benefits of drug treatment). Similarly, the Memory Component involves: (a) Memory aids (reminders and cues to be used between sessions); (b) Summarizing/reiterating information (frequent review throughout sessions); (c) Prospective memory (emphasize routine, develop cues, elaborate on positive behaviors); and (d) Environmental engineering (prepare for adverse events). Lastly, the Information Processing Component includes: (a) Mixed methods of presentation (verbal, visual, and hands-on); (b) Simple language (clear, concrete examples aligned with health literacy level); (c) Present content slowly (allow extra time for responses); and (d Immediate feedback following assessment (oral/ written).Of particular note, the investigators are using this framework to examine all combinations of these components (rather than merely testing all four) to promote ecological validity and future implementation. Specifically, our approach will help determine the most resource-efficient intervention, as there are many barriers to adding components to standard of care in these clinical settings. For example, if components targeting only two domains can produce equivalent outcomes as components targeting four, the former would be identified as preferred

ELIGIBILITY:
Inclusion Criteria:

* being 18 years or older
* meeting DSM-V criteria for opioid dependence and being newly prescribed and adherent to Medication for Opioid Use Disorder (e.g., methadone, buprenorphine) at the APT Foundation, Inc.
* showing mild cognitive impairment based on the Montreal Cognitive Assessment (MoCA) screening
* having initiated Pre-Exposure Prophylaxis (PrEP) within the past week
* confirming HIV-negative status through proof of PrEP prescription
* reporting unsafe injection drug use practices or unprotected sex within the past 3 months
* having a cell phone
* being able to read and understand in English

Exclusion Criteria:

* unable to provide consent
* actively suicidal
* actively homicidal
* actively psychotic
* display MoCA scores suggestive of dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Pre-Exposure Prophylaxis Adherence via Dried Blood Spots (DBS) | PrEP adherence DBS measured at week 4
  Dried Blood Spots will test the amount of active PrEP components in the participants blood.
Pre-Exposure Prophylaxis Adherence via Dried Blood Spots (DBS) | PrEP adherence DBS measured at the 3-month post-intervention follow-up
  Dried Blood Spots will test the amount of active PrEP components in the participants blood.
Pre-Exposure Prophylaxis Adherence via Dried Blood Spots (DBS) | PrEP adherence DBS measured at the 6-month post-intervention follow-up
  Dried Blood Spots will test the amount of active PrEP components in the participants blood.
Pre-Exposure Prophylaxis Adherence via Dried Blood Spots (DBS) | PrEP adherence DBS measured at the 9-month post-intervention follow-up
  Dried Blood Spots will test the amount of active PrEP components in the participants blood.
Pre-Exposure Prophylaxis Adherence via pharmacy refill data | PrEP adherence pharmacy refill data measured at week 4
  Pharmacy refill data confirms the participants has refilled their PrEP prescription at local pharmacy
Pre-Exposure Prophylaxis Adherence via pharmacy refill data | PrEP adherence pharmacy refill data measured at the 3-month post-intervention follow-up
  Pharmacy refill data confirms the participants has refilled their PrEP prescription at local pharmacy
Pre-Exposure Prophylaxis Adherence via pharmacy refill data | PrEP adherence pharmacy refill data measured at the 6-month post-intervention follow-up
  Pharmacy refill data confirms the participants has refilled their PrEP prescription at local pharmacy
Pre-Exposure Prophylaxis Adherence via pharmacy refill data | PrEP adherence pharmacy refill data measured at the 9-month post-intervention follow-up
  Pharmacy refill data confirms the participants has refilled their PrEP prescription at local pharmacy
Pre-Exposure Prophylaxis Adherence via self-report scale | PrEP adherence pharmacy self report measured at week 4
  Self-reported PrEP adherence is measured on a scale of 0-100, the higher the score the greater the adherence
Pre-Exposure Prophylaxis Adherence via self-report scale | PrEP adherence pharmacy self report measured at the 3-month post-intervention follow-ups
  Self-reported PrEP adherence is measured on a scale of 0-100, the higher the score the greater the adherence
Pre-Exposure Prophylaxis Adherence via self-report scale | PrEP adherence pharmacy self report measured at the 6-month post-intervention follow-ups
  Self-reported PrEP adherence is measured on a scale of 0-100, the higher the score the greater the adherence
Pre-Exposure Prophylaxis Adherence via self-report scale | PrEP adherence pharmacy self report measured at the 9-month post-intervention follow-ups
  Self-reported PrEP adherence is measured on a scale of 0-100, the higher the score the greater the adherence

SECONDARY OUTCOMES:
HIV risk behaviors questionnaire | HIV risk behaviors measured at Week 1
  Self-report of "any" high-risk behavior (sexual or drug-related) as well as measurements of event-level (i.e., partner-by-partner) behaviors.
HIV risk behaviors questionnaire | HIV risk behaviors measured at Week 4
  Self-report of "any" high-risk behavior (sexual or drug-related) as well as measurements of event-level (i.e., partner-by-partner) behaviors.
HIV risk behaviors questionnaire | HIV risk behaviors measured at the 3-month post-intervention follow-up
  Self-report of "any" high-risk behavior (sexual or drug-related) as well as measurements of event-level (i.e., partner-by-partner) behaviors.
HIV risk behaviors questionnaire | HIV risk behaviors measured at the 6-month post-intervention follow-up
  Self-report of "any" high-risk behavior (sexual or drug-related) as well as measurements of event-level (i.e., partner-by-partner) behaviors.
HIV risk behaviors questionnaire | HIV risk behaviors measured at the 9-month post-intervention follow-up
  Self-report oof "any" high-risk behavior (sexual or drug-related) as well as measurements of event-level (i.e., partner-by-partner) behaviors.
HIV prevention IMB model constructs questionnaire | HIV prevention IMB model constructs measured at Week 1
  self report of (a) information - HIV risk- and PrEP-related knowledge; (b) motivation - readiness to change and intentions to change PrEP adherence and change HIV risk behavior; (c) behavioral skills - PrEP adherence skills and HIV risk reduction skills
HIV prevention IMB model constructs questionnaire | HIV prevention IMB model constructs measured at Week 4
  self report of (a) information - HIV risk- and PrEP-related knowledge; (b) motivation - readiness to change and intentions to change PrEP adherence and change HIV risk behavior; (c) behavioral skills - PrEP adherence skills and HIV risk reduction skills
HIV prevention IMB model constructs questionnaire | HIV prevention IMB model constructs measured at the 3-month post-intervention follow-up
  self report of (a) information - HIV risk- and PrEP-related knowledge; (b) motivation - readiness to change and intentions to change PrEP adherence and change HIV risk behavior; (c) behavioral skills - PrEP adherence skills and HIV risk reduction skills
HIV prevention IMB model constructs questionnaire | HIV prevention IMB model constructs measured at the 6-month post-intervention follow-up
  self report of (a) information - HIV risk- and PrEP-related knowledge; (b) motivation - readiness to change and intentions to change PrEP adherence and change HIV risk behavior; (c) behavioral skills - PrEP adherence skills and HIV risk reduction skills
HIV prevention IMB model constructs questionnaire | HIV prevention IMB model constructs measured at the 9-month post-intervention follow-up
  self report of (a) information - HIV risk- and PrEP-related knowledge; (b) motivation - readiness to change and intentions to change PrEP adherence and change HIV risk behavior; (c) behavioral skills - PrEP adherence skills and HIV risk reduction skills

OTHER OUTCOMES:
Drug Test via Urine toxicology | conducted at Week 1
  Four-panel (i.e., heroin, cocaine, oxycodone, and benzodiazepine) immunoassay (I/A) urinalyses
Drug Test via Urine toxicology | conducted at twice weekly during the 4-week intervention phase
  Four-panel (i.e., heroin, cocaine, oxycodone, and benzodiazepine) immunoassay (I/A) urinalyses
Drug Test via Urine toxicology | conducted at 3-month follow-up
  Four-panel (i.e., heroin, cocaine, oxycodone, and benzodiazepine) immunoassay (I/A) urinalyses
Drug Test via Urine toxicology | conducted at 6-month follow-up
  Four-panel (i.e., heroin, cocaine, oxycodone, and benzodiazepine) immunoassay (I/A) urinalyses
Drug Test via Urine toxicology | conducted at 9-month follow-up
  Four-panel (i.e., heroin, cocaine, oxycodone, and benzodiazepine) immunoassay (I/A) urinalyses

CONTACTS AND LOCATIONS:
Overall Officials: Michael Copenhaver, PhD, Principal Investigator — University of Connecticut
Locations (1):
- APT Foundation, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date
Access Criteria: Proposals should be directed to Michael.Copenhaver@uconn.edu To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Mistler CB, Shrestha R, Gunstad J, Collins L, Madden L, Huedo-Medina T, Sibilio B, Copenhaver NM, Copenhaver M. Application of the multiphase optimisation strategy (MOST) to optimise HIV prevention targeting people on medication for opioid use disorder (MOUD) who have cognitive dysfunction: protocol for a MOST study. BMJ Open. 2023 Jun 30;13(6):e071688. doi: 10.1136/bmjopen-2023-071688. PMID 37399447